CLINICAL TRIAL: NCT03557450
Title: A Feasibility Study to Determine PET/CT Imaging of Blood Flow to the Bone
Acronym: PETCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1227928
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Normal Subjects
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PET/CT scanning with sodium fluoride (Experimental): Subjects will received PET/CT scanning with sodium fluoride
  Interventions: Device: PET/CT Scan

INTERVENTIONS:
Device: PET/CT Scan — PET/CT scanning with sodium fluoride

SUMMARY:
To evaluate if a commonly used medical bone scan, called positron emission tomography/computed tomography (PET/CT) with sodium fluoride can measure bone blood flow to the hip.

DETAILED DESCRIPTION:
The purpose of this research is to validate technique on a commonly used medical bone scan, called positron emission tomography/computed tomography (PET/CT) along with sodium fluoride as the tracer for determining blood flow to the bone. Up to 12 subjects will have PET/CT scans so that we can determine the repeatability and reliability of the images prior to using PET/CT for this use on subjects in the Phase 1b part of Dr. Nancy Lane's clinical research study entitled "A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study of the Safety and Tolerability of Intravenous LLP2A-Alendronate in Adult Men and Women with Osteopenia Secondary to Glucocorticoids" (IRB Protocol #866350).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study.

1. 20 - 75 years old
2. Must be ambulatory and able to attend all appointments
3. Women must agree to use one of the following methods of birth control for the duration of the clinical trial:

   systemic hormonal contraceptive (oral, injected, transdermal), intrauterine device, double barrier (e.g., cervical cap or diaphragm with condom or spermicide). Men with female partners must agree to use double barrier contraception, unless their partner is using systemic hormonal contraceptives or has an intrauterine device
4. Subject undergoing PET/CT scans must have the ability to lay motionless for up to 30 minutes.

Exclusion Criteria:

1. Subjects undergoing PET/CT scans must not be breast-feeding.
2. History of hypersensitivity to fluoride

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Measure of Blood Flow to the proximal femur | Within a week of the scan
  Measure the sodium fluoride -18 concentration to blood vessels of the the proximal femur

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No